CLINICAL TRIAL: NCT05529043
Title: MINISTOP Plus Program for Pre-school Children With Overweight and Obesity: A Pilot Randomized Controlled Trial
Brief Title: MINISTOP Plus Program for Pre-school Children With Overweight and Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christine Delisle Nyström, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-02956-01
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINISTOP app (Active Comparator): Receives the MINISTOP app for 12-months.
  Interventions: Behavioral: MINISTOP app
- MINISTOP Plus Program (Experimental): Receives the MINISTOP app for 12-months and receives Community Group Mini.
  Interventions: Behavioral: MINISTOP Plus Program

INTERVENTIONS:
Behavioral: MINISTOP app — The MINISTOP app is a behavioural change program aiming to promote healthier diet and physical activity behaviours in pre-school children. The program consists of features such as information, monitoring and feedback (dietary variables, physical activity, and screen time) and it is built around 13 themes. The participants will have access to the app for 12-months.
  Arms: MINISTOP app
Behavioral: MINISTOP Plus Program — Consists of the MINISTOP app and the Community Group Mini. The Community Group Mini consists of group activities to promote physical activity for both children and parents. The Community Group Mini will meet once per week in different playgrounds and nature reserves and will be organized by a trained group leader.
  Arms: MINISTOP Plus Program

SUMMARY:
The Mobile-based intervention intended to stop obesity in preschoolers (MINISTOP) program has been developed to be a comprehensive digital support program for all children irrespective of weight status. However, a one size fits all approach may not be sufficient as some families may require extra support through in-person activities to achieve the required lifestyle behaviour change in order to attain and maintain a healthy weight. Therefore, the aims of this pilot randomized controlled trial are to evaluate the efficacy and feasibility of the MINISTOP Plus Program in pre-school children with overweight and obesity on: (i) children's BMI z-scores; (ii) intake of fruit and vegetables, sweet and savoury snacks, and sweet drinks; (iii) time spent in different physical activity intensities; (iv) screen time; and (v) parental self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 5 year old children with overweight and obesity residing in the municipality of Kungsbacka.

Exclusion Criteria:

* If a child has a disease or disorder that affects body size or feeding.
* Children who have a parent suffering from a serious physical or psychological disease making the study too demanding for the family.
* Children from families who will not be able to understand the app content, i.e., those who do not speak Swedish, English, Arabic, or Somali

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Body mass index | At the end of the intervention which is 12-months after baseline
  Body weight divided by height squared

SECONDARY OUTCOMES:
Intake of key dietary indicators as assessed by a questionnaire. | At the end of the intervention which is 12-months after baseline.
  Intake of fruits, vegetables, sweet snacks, savoury snacks, and sweet drinks (grams/day)
Physical activity assessed using an accelerometer | At the end of the intervention which is 12-months after baseline
  Time spent in different physical activity intensities, i.e., sedentary, light, moderate, vigourous, and moderate-to-vigorous physical activity (minutes/day)
Screen time as assessed by a questionnaire | At the end of the intervention which is 12-months after baseline
  Number of minutes per day spent in front of a screen
Self-efficacy self-efficacy for promoting healthy dietary and physical activity behaviours in their children's | At the end of the intervention which is 12-months after baseline
  Questionnaire to parents

CONTACTS AND LOCATIONS:
Overall Officials: Christine Delisle Nyström, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Biosciences and Nutrition, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No